CLINICAL TRIAL: NCT06747351
Title: A Phase 3, Single-Arm, Multiple-Dose, Pharmacokinetic Comparability Trial Between TAK-881 and HYQVIA in Adults With Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Brief Title: A Study to Compare TAK-881 and HYQVIA in Adults With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-881-3003; 2024-517450-95-00 (EU CTIS Number); jRCT2041250014 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Keywords: Immunoglobulin; facilitated subcutaneous , Immunoglobulin;; Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All Participants (HYQVIA and TAK-881) (Experimental): Ramp-up Epoch:
  Participants on IGIV or cIGSC will switch to HYQVIA during ramp-up epoch with gradually increasing doses/volumes. For participants switching from IGIV, first HYQVIA dose is given two weeks after their last IGIV infusion. For participants switching from cIGSC, first dose is given one week after a weekly infusion or two weeks after a bi-weekly infusion, using a SC investigational needle set.
  Treatment Epoch:
  After completing ramp-up, participants will enter HYQVIA dosing epoch 2-3 weeks later, depending on treatment interval. Those already on HYQVIA at screening will skip ramp-up and proceed directly to dosing phase, lasting 18 weeks for a 3-week interval and 20 weeks for 4-week interval. After HYQVIA PK sampling period, participants will switch to TAK-881 with a 1:1 dose conversion. TAK-881 dosing lasts 24 weeks with a SC infusion needle set.
  Extension Epoch:
  Post-TAK-881, participants will enter the extension epoch, continuing treatment for up to 3 years.
  Interventions: Biological: TAK-881; Biological: HYQVIA; Device: SC Investigational Needle Sets

INTERVENTIONS:
Biological: TAK-881 — Participants will receive SC infusion of TAK-881.
  Other Names: Immune Globulin Subcutaneous (Human); 20% Solution with Recombinant Human Hyaluronidase (rHuPH20).
Biological: HYQVIA — Participants will receive SC infusion of HYQVIA.
  Other Names: Immune Globulin Infusion (Human); 10% Solution with rHuPH20
Device: SC Investigational Needle Sets — The single-use only SC needle set will be used to administer TAK-881/HYQVIA to the target depth below the skin surface. One needle set (single or bifurcated) will be used per infusion.

SUMMARY:
The main aim of this study is to evaluate the pharmacokinetic (PK) comparability between TAK-881 and HYQVIA subcutaneous (SC) administration for maintenance therapy of CIDP.

The participants who are already receiving intravenous immunoglobulin G (IGIV), conventional subcutaneous intravenous immunoglobulin G (cIGSC), or HYQVIA will be treated with the same dose equivalent as their prior IG treatment with HYQVIA for 20 weeks followed by TAK-881 for 24 weeks.

Participants will need to visit the clinic every 3 or 4 weeks until they enter the extension phase. In the extension phase, home infusions are allowed, and visits will occur between every 12 weeks and 24 weeks.

DETAILED DESCRIPTION:
The study includes a screening phase, a ramp-up phase (if needed), a HYQVIA treatment phase, a TAK-881 treatment phase, and an extension phase. Participants who have been receiving cIGSC or IGIV prior to the study will enter a HYQVIA ramp-up phase, starting 1 to 2 weeks after their last pre-study cIGSC or IGIV dose. Participants already on HYQVIA at the time of screening will proceed directly to the treatment phase. After the TAK-881 dosing phase, participants will move on to the TAK-881 extension phase, with the preference for subsequent infusions in the extension phase to be administered by the participant or caregiver at home.

ELIGIBILITY:
Inclusion Criteria

* Participant is willing and able to understand and fully comply with trial procedures and requirements, in the opinion of the investigator.
* Participant has provided informed consent (that is, in writing, documented via a signed and dated informed consent Form [ICF]) and any required privacy authorization before the initiation of any trial procedures.
* Participant has a documented diagnosis of CIDP or possible CIDP, as confirmed by a neurologist specializing/experienced in neuromuscular diseases and consistent with the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) 2021 criteria.
* Participant has responded to IgG treatment in the past (documented partial or complete resolution of neurological symptoms and deficits).
* Participant is on a stable, pretrial treatment with IGIV, cIGSC, or HYQVIA (also known as TAK-771 in Japan) within the dose range equivalent to a cumulative monthly IgG dose of 0.4 to 2.4 grams per kilogram (g/kg) body weight (BW) (inclusive) administered for at least 12 weeks before screening. The dosing interval of IGIV treatment must be between 2 and 6 weeks (inclusive). The dosing interval must be weekly or biweekly for cIGSC dosing and less than or equal (<=) to 6 weeks for HYQVIA dosing. Prior to screening, variations in the dosing interval of up to +-7 days or monthly dose amount of up to +-20 percentage (%) between the participant's pretrial IgG infusions are acceptable.
* Participant has an INCAT disability score between 0 and 7 (inclusive). Participants will be eligible if one of the below eligibility criteria are met:

  1. Screening INCAT disability score of between 3 and 7 inclusive.
  2. Screening INCAT disability score of 2 (both points are from lower extremities).
  3. Screening INCAT disability score of 2 (both points are not from lower extremities) AND has at least a score of 2 or greater documented in the medical record before screening. If a score was greater than 2 documented in the medical record before screening at least 2 points must be from lower extremities.
  4. Screening INCAT disability score of 0 or 1 AND has at least a score of 2 or greater (both from lower extremities) documented in the medical record before screening, at least 2 points must be from lower extremities.
* If a participant has the potential to become pregnant, they must have a negative pregnancy test at screening and agree to employ a highly effective contraceptive measure throughout the course of the trial and for at least 30 days after the last administration of the investigational medical product (IMP).

Exclusion Criteria

* Participant with documented diagnosis of focal, multifocal, distal, or sensory CIDP, or possible focal, multifocal, distal, or sensory CIDP per the EFNS/PNS 2021 criteria.
* Participant has any neuropathy of other causes, including:

  1. Hereditary demyelinating neuropathies, such as hereditary sensory and motor neuropathy (HSMN), Charcot-Marie-Tooth (CMT) disease, and hereditary sensory and autonomic neuropathies (HSANs).
  2. Neuropathies secondary to infections, disorders, or systemic diseases such as Borrelia burgdorferi infection (Lyme disease), diphtheria, systemic lupus erythematosus, POEMS (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes) syndrome, osteosclerotic myeloma, diabetic and non-diabetic lumbosacral radiculoplexus neuropathy, lymphoma, amyloidosis.
  3. Multifocal motor neuropathy (MMN).
  4. Drug, biologic, chemotherapy, or toxin-induced peripheral neuropathy.
* Participant has any chronic or debilitating disease, or central nervous disorder that causes neurological symptoms or which may interfere with assessment of CIDP or outcome measures, including (but not limited to) multiple sclerosis, arthritis, stroke, Parkinson's disease, and diabetic peripheral neuropathy.

Note: Participants with clinically diagnosed diabetes mellitus who do not have diabetic peripheral neuropathy and who have adequate glycemic control with hemoglobin A1c [HbA1c] level of less than (<) 7.5% at screening will be eligible for the trial, provided the electrodiagnostic criteria are consistent with the diagnosis of CIDP or possible CIDP consistent with the EFNS/PNS 2021 criteria and the participant agrees to maintain adequate glycemic control.

* Participant is required to take or has taken immunomodulatory/immunosuppressive agents (except IGIV, cIGSC, or fIGSC) that include but are not limited to specific complement inhibitors, rituximab, neonatal FC receptor inhibitors (e.g. efgartigimod), and chemotherapeutic drugs, within 6 months of screening.
* Participant is required to take or has taken long-term systemic corticosteroids defined as dosages greater than (>) 20 milligrams per day (mg/day) prednisone-equivalent for >30 days within 3 months of screening.

Note: Participants using short-pulse dose corticosteroid course and oral daily corticosteroids <= 20 mg/day prednisone-equivalent are allowed.

* Participant has undergone plasma exchange within 3 months before screening.
* Participant has immunoglobulin M (IgM) paraproteinemia, including IgM monoclonal gammopathy with a high titer of antibody to myelin-associated glycoprotein.
* Participant has immunoglobulin A (IgA) deficiency (IgA <0.07 grams per liter [g/L]) associated with known anti-IgA antibodies and a history of hypersensitivity to human immunoglobulin treatment.
* Participant has a condition(s) which could alter protein catabolism and/or IgG use (for example [eg.] protein losing enteropathies, and nephrotic syndrome).
* Participant has a history or clinical manifestations of chronic kidney disease, or glomerular filtration rate of <30 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) estimated based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at the time of screening.
* Participant has a history of malignancy with less than 2 years of complete remission before screening, or active malignancy requiring chemotherapy and/or radiotherapy.

Note: Participants with adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or stable prostate cancer not requiring treatment are eligible.

* Participant has congestive heart failure (New York Heart Association class III/IV), unstable angina, unstable cardiac arrhythmias, or uncontrolled hypertension (defined as diastolic blood pressure >100 millimeters of mercury (mm Hg) and/or systolic blood pressure >160 mm Hg during the screening epoch confirmed on 2 measures >30 minutes apart).
* Participant has an acquired or inherited thrombophilic disorder, such as protein C deficiency, protein S deficiency, antithrombin deficiency, and primary antiphospholipid antibody syndrome.
* Participant has a history of deep vein thrombosis or arterial thromboembolic events (eg, cerebrovascular accident, pulmonary embolism) within 12 months before screening.
* Participant has any medical condition, laboratory finding, or physical examination finding that precludes participation or with clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may interfere with successful completion of the trial or place the participant at undue medical risk.
* Participant has a known history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following IGIV, IGSC, and/or immune serum globulin infusions.
* Participant has a known systemic hypersensitivity to any of the excipients of TAK-881/HYQVIA in accordance with the Investigator's Brochure (IB)/package insert/Summary of Product Characteristics (SmPC).
* Participant has a known systemic hypersensitivity to hyaluronidase or rHuPH20.
* Participant has a known history of positive result for or is positive at screening for one or more of the following: hepatitis B surface antigen (HBsAg), polymerase chain reaction (PCR) for hepatitis C virus (HCV), PCR for Human Immunodeficiency Virus (HIV) Type 1 and Type 2.

Note: Cured participants with a history of hepatitis C infection who have a negative PCR test at screening are eligible.

* Participant has clinically significant anemia that precludes repeated blood sampling during the trial, or hemoglobin level of <10.0 grams per deciliter (g/dL) at the time of screening.
* Participant has any of the following laboratory values at screening:

  1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2.5*upper limit of normal (ULN).
  2. Platelet count <100,000 cells per microliter (cells/µL).
  3. Absolute neutrophil count <1000 cells/µL.
* If female, the participant is pregnant or lactating at the time of screening.
* Participant has participated in another clinical trial involving an IMP or investigational device within 12 weeks or 5 half-lives, whichever is longer, before enrollment (except for participants rolling over from the Japan study TAK-771-3002) or is scheduled to participate in another clinical trial involving an IMP or investigational device during the course of this trial.
* Participant is a trial site employee, an immediate family member (eg, spouse, parent, child, sibling), or is in a dependent relationship with a trial site employee who is involved in conduct of this trial or may consent under duress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2028-06-25 (Estimated); Study Completion 2028-06-25 (Estimated)

PRIMARY OUTCOMES:
Baseline-Uncorrected Area Under the Curve During the Dosing Interval at Steady-State (AUC0-tau;ss) Based on Total Immunoglobulin G (IgG) Levels | 3-Week dosing: Day 1 (pre- and post-infusion), 24, 72, 120 hours and 7, 14, 17, 21 days (post-infusion); 4-Week dosing: Day 1 (pre- and post-infusion), 24, 72, 120 hours and 7, 14, 21, 28 days (post-infusion) of last infusion

SECONDARY OUTCOMES:
Baseline-Uncorrected Area Under the Curve to the Last Measurable Concentration at Steady-State (AUClast,ss) Based on Total IgG Levels | 3-Week dosing: Day 1 (pre- and post-infusion), 24, 72, 120 hours and 7, 14, 17, 21 days (post-infusion); 4-Week dosing: Day 1 (pre- and post-infusion), 24, 72, 120 hours and 7, 14, 21, 28 days (post-infusion) of last infusion
Baseline-Uncorrected Time of the Last Measurable Concentration at Steady-State (Tlast,ss) Based on Total IgG Levels | 3-Week dosing: Day 1 (pre- and post-infusion), 24, 72, 120 hours and 7, 14, 17, 21 days (post-infusion); 4-Week dosing: Day 1 (pre- and post-infusion), 24, 72, 120 hours and 7, 14, 21, 28 days (post-infusion) of last infusion
Baseline-Uncorrected Maximum Observed Concentration at Steady-State (Cmax,ss) Based on Total IgG Levels | 3-Week dosing: Day 1 (pre- and post-infusion), 24, 72, 120 hours and 7, 14, 17, 21 days (post-infusion); 4-Week dosing: Day 1 (pre- and post-infusion), 24, 72, 120 hours and 7, 14, 21, 28 days (post-infusion) of last infusion
Baseline-Uncorrected Time to Maximum Concentration at Steady-State (Tmax,ss) Based on Total IgG Levels | 3-Week dosing: Day 1 (pre- and post-infusion), 24, 72, 120 hours and 7, 14, 17, 21 days (post-infusion); 4-Week dosing: Day 1 (pre- and post-infusion), 24, 72, 120 hours and 7, 14, 21, 28 days (post-infusion) of last infusion
Total IgG Trough Level | Up to 4.06 years
Number of Participants With Adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) who Experienced Relapse Related to Baseline | Baseline up to 24 weeks
  Relapse is defined as an increase in the adjusted INCAT disability score by greater than and equal to (>=) 1-point relative to the baseline score. The INCAT disability score is a clinician-reported measure of a participant's level of arm and leg impairment. The arm and leg components of the INCAT are scored between 0 and 5 points (where arm = 0 indicates 'no upper limb problems' and arm = 5 indicates 'inability to use either arm for any purposeful movement', and leg = 0 indicates 'walking not affected', and leg = 5 indicates 'restricted to wheelchair, unable to stand and walk a few steps with help') and are summed to produce the overall INCAT disability score ranging between 0 and 10 points. A score of 0 indicates no signs of disability) and 10 indicates the most severe disability.
Change From Baseline in Hand Grip Strength | Baseline up to 24 weeks
  Grip strength assessments conducted by prescribing physicians using the Martin Vigorimeter or the Jamar Dynamometer (as available at the site and performed per routine clinical practice).
Change From Baseline in Medical Research Council (MRC) Sum Score | Baseline up to 24 weeks
  The MRC sum score measures muscle strength from both the left and right sides of the body on a scale of 0 to 5. The total MRC sum score ranges from 0 (paralysis) to 60 (normal strength), where higher score indicates better strength.
Change From Baseline in Inflammatory Rasch-built Overall Disability Scale (I-RODS) Centile Score | Baseline up to 24 weeks
  The I-RODS is a validated, participants self-reported, linearly weighted overall disability scale that was specifically designed to capture current activity and social participation limitations in participants with immune-mediated peripheral neuropathies including CIDP. The I-RODS comprises 24 items for which participants are asked to rate their functioning related to a variety of everyday tasks at the moment of completion. The participant assigns a score between 0 and 2 to each item as follows: 0 (impossible to perform), 1 (performed with difficulty), 2 (easily performed) with a lower score indicating more severe activity and social participation limitations.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to 4.06 years
Number of Participants With Infusion Withdrawals, Interruptions, and Infusion Rate Reductions due to TAK-881-related TEAEs | Up to Week 55
Number of Participants With Positive Binding Antibodies (Titer Greater than and equal to [>=] 1:160) and With Positive Neutralizing Antibodies to rHuPH20 | Up to 4.06 years
Number of Infusions per Month at Full Dose With Both TAK-881 and HYQVIA in all Participants | Up to 4.06 years
Number of Infusions Sites (Needle Sticks) per Month at Full Dose With Both TAK-881 and HYQVIA in all Participant | Up to 4.06 years
Number of Infusions Sites (Needle Sticks) per Infusion at Full Dose With Both TAK-881 and HYQVIA in all Participants | Up to Week 55
Duration of Infusions (Minutes) at Full Dose With Both TAK-881 and HYQVIA in all Participants | Up to 4.06 years
Monthly Infusion Time (Minutes/Month) at Full Dose With Both TAK-881 and HYQVIA in all Participants | Up to 4.06 years
Maximum Tolerated Infusion Rate per Site (milliliter [mL]/hour/site) at Full Dose With Both TAK-881 and HYQVIA in all Participants | Up to Week 55
Infusion Volume per Site (mL/site) at Full Dose With Both TAK-881 and HYQVIA in all Participants | Up to Week 55
Time of Infusion Preparation Measured by Healthcare provider (HCP) | Up to 4.06 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (52):
- United States (16):
  - HonorHealth Neurology, Scottsdale, Arizona
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Neurology Associates, Maitland, Florida
  - Knight Neurology, Rockledge, Florida
  - The Washington University, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - University of North Carolina (UNC), Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University (OHSU) - Nephrology and Hypertension Clinic - Marquam Hill, Portland, Oregon
  - Neurology Rare Disease Center, Denton, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - BCN Research, LLC, Greenfield, Wisconsin
- Argentina (2):
  - INECO, Rosario, Santa Fe Province
  - Instituto Argentino de Investigacion Neurologica (IADIN), Buenos Aires
- Fakultni nemocnice Hradec Kralove, Hradec Králové, Czechia
- Denmark (2):
  - Copenhagen University Hospital, Copenhagen, Capital Region
  - Aarhus Universitetshospital, Aarhus, Central Jutland
- Germany (5):
  - Universitätsklinikum Mannheim GmbH, Mannheim, Baden-Wurttemberg
  - University of Ulm, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Marburg, Marburg, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Charite - Universitatsmedizin Berlin, Berlin
- Greece (2):
  - Attikon University General Hospital, Athens, Attica
  - University General Hospital of Patras, Patras, Peloponnese
- Italy (9):
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan, Lombardy
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano, Lombardia
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano, Torino, Piemonte
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia, Brescia
  - Ospedale San Martino, Genova
  - Az Ospedaliera Universitaria Policlinico G Martino, Messina
  - Fondazione Istituto Neurologico Casimiro Mondino, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
- Japan (8):
  - Japan Organization of Occupational Health and Safety Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Tohoku Medical and Pharmaceutical University Hospital, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara, Nara
  - Higashimatsuyama Municipal Hospital, Higashi-Matsuyama, Saitama
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Tokushima University Hospital, Tokushima, Tokuchima
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
- Poland (4):
  - Oddzial Kliniczny Neurologii, Krakow, Lesser Poland Voivodeship
  - Clinirem Sp zo.o., Lublin, Lublin Voivodeship
  - Warszawski Uniwersytet Medyczny, Warsaw, Masovian Voivodeship
  - Copernicus Podmiot Leczniczy, Gdansk, Pomeranian Voivodeship
- Spain (2):
  - Hospital de La Santa Creu I San Pau, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/b6cac22e9fdf4adc??page=1&idFilter=TAK-881-3003